CLINICAL TRIAL: NCT05119504
Title: Improving the Experience of Exercise Among Individuals With Internalized Weight Bias Using Acceptance-based Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: The Obesity Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1689962
Record Dates: First submitted 2021-11-01; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals conducting study assessments will remain masked to treatment condition.
  Interventions have been matched for time, so that masked assessors are unable to note a discrepancy in treatment condition throughout study procedures. Intervention staff will be responsible for preparing the room with materials and for relocating participant from intervention room back to the assessment room so that the masked assessor is not able to view any materials left behind from the treatment condition. Participants will be reminded by study staff throughout study procedures that they should not disclose their treatment condition or information about their intervention meeting that could inform masked staff of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance-based (Experimental): This 90-minute one-on-one intervention will provide psychoeducation and experiential training on the use of acceptance-based strategies for physical activity.
  Interventions: Behavioral: Acceptance and Commitment
- Multi Health Behavior (Sham Comparator): This 90-minute one-on-one intervention will provide psychoeducation on physical activity as one of several interconnected health behaviors.
  Interventions: Behavioral: Multi-Health Behavior

INTERVENTIONS:
Behavioral: Acceptance and Commitment — During the 90-minute, one-on-one interventionist led session, participants will learn three inter-related acceptance-based techniques tailored for coping with physical discomfort and negative affect during physical activity. (1) cognitive defusion (i.e., disentangling physical sensations and thoughts from behavior), (2) acceptance (i.e., increasing willingness to experience unpleasant physical sensations/negative affect without trying to change or control them), and (3) valued action (i.e., evaluating the role of physical activity as a valued behavior). Participants will be taught these techniques via didactic instruction, metaphors, and experiential activities.
  All participants will receive a two-week physical activity prescription based on national guidelines recommending 150 minutes of at least moderate intensity physical activity per week.
  Arms: Acceptance-based
Behavioral: Multi-Health Behavior — The multi health behavior condition will include didactic material focused broadly on healthy lifestyle recommendations including physical activity. It will also emphasize that physical activity is one of several interconnected health behaviors including balanced diet, sleep, stress management. All participants will receive a two-week physical activity prescription based on national guidelines recommending 150 minutes of at least moderate intensity physical activity per week.
  Arms: Multi Health Behavior

SUMMARY:
The goal of this study is to test whether an acceptance based intervention can modify the relationship between heart rate and perceived exertion/negative during physical activity among individuals who have a high degree of internalized weight bias.

DETAILED DESCRIPTION:
In this two-phase pilot, we will first test in a controlled setting whether an acceptance-based intervention can modify the relationship between Heart Rate and perceived exertion/negative affect during moderate intensity physical activity among individuals high in internalized weight bias (Phase 1) and then evaluate these mechanisms in real-time during uptake of a two-week physical activity prescription (Phase 2). Using a 2x2 factorial design, we will randomize individuals with Body Mass Index (BMI) ≥25, high and low internalized weight bias, and insufficient activity (<60 min of moderate physical activity/week) to receive a 90-minute acceptance-based intervention workshop versus a multi-health behavior education condition prior to completing a 30-minute session of supervised, moderate intensity treadmill walking. Heart rate, self-reported perceived exertion and affect will be assessed throughout physical activity.

For Phase 2, all participants from Phase 1 will receive a two-week physical activity prescription consistent with National Guidelines (150 minutes moderate intensity aerobic physical activity, recommended in 30-minute bouts) to determine the effect of treatment condition on subsequent adherence to physical activity. Physical activity adherence will be monitored with Actigraphy and Ecological Momentary Assessment (repeated daily surveys via smartphone) will be used to evaluate participant self-efficacy, intention, motivation for physical activity in near real-time.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old,
* BMI 25-40 kg/m2
* insufficiently active (<60 minutes of moderate intensity activity per week).
* High/low internalized weight bias
* Access to personal smartphone device and willing to download free smartphone app for data collection

Exclusion Criteria:

* Comorbid issues that might interfere with ability to engage in physical activity
* Factors that would influence ability to complete study protocol (e.g., cognitive, psychological)
* medication that would affect heart rate (e.g., beta blocker),
* women who are nursing or pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in perceived exertion | Every five minutes during 30-minute treadmill session
  Assessed using the Borg Ratings of Perceived Exertion-Participants are prompted verbally to rate their exertion on a scale ranging from 6 (no exertion at all) to 20 (maximum exertion) every 5 minutes.
Change in affect | Every five minutes during 30-minute treadmill session
  Assessed using the Feeling Scale --This single-item measure assesses how participants feel 'at the present moment' on an 11-point scale ranging from -5 (very bad) to +5 (very good)), administered every 5 minutes during PA

SECONDARY OUTCOMES:
Physical Activity Adherence | Daily for 14 days
  For two weeks following the intervention condition, physical activity will be objectively measured using the ActiGraph GT9X Link. This device, worn on the non-dominant wrist, has been previously validated to assess movement and associated energy expenditure. Minute-by-minute data will be analyzed to determine the amount of time spent in bout-related moderate intensity PA (≥ 3 METs, ≥10 min), metrics to increase the likelihood of capturing 'purposeful' PA
Exercise self-efficacy, intention, motivation | Four times per day for 14 days
  Using the Lifedata platform which includes the RealLife EXP application that can be downloaded onto participants' smartphones, participants will be prompted via vibration and audible tone to complete EMA surveys on self-efficacy, intention, and motivation for PA. Items are adapted from validated measures used in the physical activity literature. Participants will be prompted to complete a survey semi-randomly near four anchor times throughout the day, with 90 minutes to respond.

CONTACTS AND LOCATIONS:
Overall Officials: KayLoni Olson, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
Consistent with Lifespan IRB policy, any interested individuals seeking access to conduct secondary analysis of study data will be required to submit a formal agreement with the PI, or designee, that 1) the data will be used for research purposes only and will not be used to identify any individual participants, 2) the data will be secured using appropriate computer technology, and 3) that the data will be destroyed or returned to the PI after the analyses are complete. This will be mediated by IRB involvement and the PI retains the right to deny any request for qualitative data access.
  Generally, we work with the requestor/user to provide the minimum data necessary for their research question to support resource sharing while maintaining patient confidentiality.